CLINICAL TRIAL: NCT00327626
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Activity of ISIS 113715 Administered Daily in Patients With Type 2 Diabetes Mellitus Being Treated With Sulfonylurea
Brief Title: Safety, Tolerability, and Activity of ISIS 113715 in People With Type 2 Diabetes Mellitus Being Treated With Sulfonylurea
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study was never started due to regional geopolitical conflict
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 113715-CS12
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2007-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Fasting plasma glucose; HbA1c; Oral antidiabetic agent(s)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ISIS-113715

INTERVENTIONS:
Drug: ISIS 113715

SUMMARY:
The aim of this study is to evaluate the safety, tolerability, and pharmacokinetics of two ISIS 113715 subcutaneous doses (15 mg and 30 mg/day) in combination with oral antidiabetic agents (OAD) versus OAD + placebo in patients with inadequately controlled type 2 diabetes, despite ongoing maximal treatment with OAD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (post-menopausal and/or surgically sterile)
* Aged 18 to 70 years
* Diagnosed with type 2 diabetes mellitus of eight years or less in duration
* Being treated with OAD at stable maximum doses [defined as at least 10 mg/day glibenclamide (preferred), or 20 mg/day glipizide, with or without at least 1,500 mg/day metformin] for at least three months prior to screening
* Having fasting plasma glucose levels of 150-270 mg/dL and HbA1c levels of 7.5-11.0%

Exclusion Criteria:

* Greater than 3 severe hypoglycemic episodes within six months of screen
* Pregnant, breastfeeding, or intends to become pregnant
* Clinical signs or symptoms of liver disease, acute, or chronic hepatitis, or ALT greater than the upper limit of normal
* Positive hepatitis B surface antigen, hepatitis C antibody, or HIV test
* Patients with history of renal transplantation or renal dialysis or microalbuminuria defined as urine albumin > 200 mg/day
* History of insulin use within three months of screen
* History of diabetic ketoacidosis
* Treatment with any thiazolidinedione (e.g., rosiglitazone) within three months of screen
* History of lactic acidosis while on metformin therapy
* Complications of diabetes (e.g., neuropathy, nephropathy, and retinopathy)
* Clinically significant and currently active diseases
* Clinical significant abnormalities in medical history, physical examination, or laboratory examination

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2007-02-01 (Actual); Study Completion 2007-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety, tolerability, and pharmacokinetics of two ISIS 113715 subcutaneous dosages in combination with OAD versus OAD + placebo.
Examine the effect of treatment with 15 and 30 mg/day ISIS 113715 on fasting plasma glucose and HbA1c.
Evaluate the effects of ISIS 113715 on insulin sensitivity, B-cell function, proinsulin/insulin ratio, fasting insulin, C-peptide and proinsulin.

CONTACTS AND LOCATIONS:
Overall Officials: Mark K Wedel, MD, JD, FACP, Study Director — Ionis Pharmaceuticals, Inc.
Locations (5):
- Israel (5):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Western Galilee Medical Center - Nahariya, Nahariya
  - Kaplan Medical Center, Rehovot
  - ZIV Hospital, Safed